CLINICAL TRIAL: NCT07347301
Title: 30-Day Postoperative Infection Rate in Pediatric Tonsillectomy: Head-Drape vs. Full-Body Surgical Draping
Brief Title: Head-Only Draping in Pediatric Tonsillectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-01372
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Tonsillectomy; Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Head-Only Draping (Experimental): Pediatric tonsillectomy will be performed with head-only draping.
  Interventions: Other: Head-Only Surgical Draping
- Full-Body Draping (Active Comparator): Pediatric tonsillectomy will be performed with traditional full-body draping.
  Interventions: Other: Full-Body Surgical Draping

INTERVENTIONS:
Other: Full-Body Surgical Draping — Standard full-body drape.
  Arms: Full-Body Draping
Other: Head-Only Surgical Draping — Use of head drape instead of full-body drape.
  Arms: Head-Only Draping

SUMMARY:
This single-center, interventional study will compare 30-day postoperative infection rates in pediatric tonsillectomy performed with either head-only draping or traditional full-body draping. Secondary analyses will evaluate differences in waste production, material and disposal costs, and provider attitudes between the two draping techniques. This study will randomize participants 1:1 to either the head-only draping cohort (intervention) or the full-body draping cohort (control).

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients <18 years at time of surgery.
2. Scheduled for tonsillectomy, with or without adenoidectomy, without any other procedures requiring full-body draping.
3. Ability to complete 30-day outcome assessment (i.e., remain in follow-up or reachable via phone/electronic health record).
4. Parent/guardian able to provide parental permission and consent for both them and their children.

Exclusion Criteria:

1. Significant deviation from planned surgical technique during case.
2. Pre-existing systemic infection prior to surgery.
3. Known immunodeficiency or current systemic immunosuppressive therapy.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
30-day postoperative infection rate | Day 30 Post Operation

SECONDARY OUTCOMES:
Total weight of waste | Day 0 (Day of Operation)
Disposal costs | Day 0 (Day of Operation)

CONTACTS AND LOCATIONS:
Overall Officials: Neelima Tummala, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: neelima.tummala@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to neelima.tummala@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.